CLINICAL TRIAL: NCT03787511
Title: Chronic Cough and Small Fiber Neuropathy
Acronym: CHROCOS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: patients difficult to recruit
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RC31/18/0423; 2018-A03340-55 (Other: ID-RCB)
Record Dates: First submitted 2018-12-21; First posted 2018-12-26 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Chronic Cough; Type 2 Diabetes
Keywords: cough; diabetes; small fiber neuropathy
MeSH Terms: conditions — Chronic Cough; Diabetes Mellitus, Type 2; Cough; Diabetes Mellitus; Small Fiber Neuropathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Diabetic patients with chronic cough (Other): Diabetic patients with chronic cough defined by cough lasting for more than 8 weeks. Cough assessment, neurological tests and cardiovascular tests and skin biopsy.
  Interventions: Other: Cough assessment; Other: Neurological tests and cardiovascular tests; Other: Skin biopsy
- Diabetic patients without chronic cough (Other): Diabetic patients without chronic cough defined by cough lasting for more than 8 weeks. Cough assessment, neurological tests and cardiovascular tests and skin biopsy.
  Interventions: Other: Cough assessment; Other: Neurological tests and cardiovascular tests; Other: Skin biopsy

INTERVENTIONS:
Other: Cough assessment — Cough assessment with cough visual analog scale (VAS), and Leicester Cough Questionnaire (LCQ) for Diabetic patients with chronic cough and Diabetic patients without chronic cough
Other: Neurological tests and cardiovascular tests — Neurological tests : electromyography, thermotest, QSAR + cardiovascular test for Diabetic patients with chronic cough and Diabetic patients without chronic cough
Other: Skin biopsy — Skin biopsy to evaluate small fiber neuropathy for Diabetic patients with chronic cough and Diabetic patients without chronic cough

SUMMARY:
Diabetic patients with and without chronic cough will be included in this study. After giving their informed consent, the patients will perform a spirometry, chest X-ray at the inclusion visit. Cough will be assessed using the cough visual analog scale (VAS) and the Leicester Cough Questionnaire (LCQ). Within 60 days, the patient will perform neurophysiological tests. The neurophysiological assessment will be concluded with a skin biopsy to evaluate small fiber neuropathy. The aim of the study is to compare the proportion of small fiber neuropathy between diabetic patients with chronic cough and those without chronic cough.

DETAILED DESCRIPTION:
Chronic cough is a very common entity that affects 9.6% people worldwide. Given the high number of patients with refractory cough, the concept of cough hypersensitivity syndrome (CHS) has emerged. In CHS, afferent sensory nerves may exhibit a modification of activation patterns with facilitation of encoding signals in response to irritating stimuli. Similar patterns with neuropathic pain have been described. Small fiber neuropathy has never been assessed in chronic cough. Interestingly, diabetic patients experienced cough more frequently than healthy subject. We hypothesized that small fiber neuropathy may explain chronic cough is more frequent in diabetic patients.

Within 60 days after inclusion, diabetic patients with and without chronic cough will perform neurophysiological tests such as electromyography, thermotest, QSART (Quantitative Sudomotor Axon Reflex Test and Sudoscan), cardio-vascular tests to study the autonomic nervous system. No risks are expecting with these non-invasive tests. A skin biopsy to evaluate small fiber neuropathy will also be performed.After the neurophysiological tests, a consultation will be scheduled at 6 months. A cough VAS and LCQ will be used to assess cough.

ELIGIBILITY:
Inclusion Criteria:

In diabetic patients with chronic cough:

* Chronic cough defined by cough for more than 8 weeks.
* Normal chest X-ray
* history of type 2 diabetes
* Age of diabetes onset> 40 years
* Affiliated or beneficiary person of social security
* Free, informed and written consent

In diabetic patients without chronic cough

* History of type 2 diabetes
* Age of discovery of diabetes> 40 years
* Affiliated or beneficiary person of social security
* Free, informed and written consent

Exclusion Criteria:

* Presence of physical signs of peripheral neuropathy
* Active smoking or smoking cessation within the last 12 months
* Pregnant or lactating woman
* History of non-type 2 diabetes (type I, secondary diabetes, monogenic ...)
* Cancer within the last 5 years (except cutaneous squamous cell carcinoma)
* History of anti-cancer chemotherapy
* Suspicion of autoimmune pathology
* Active neurological pathology
* Electromyography in favor of large fiber neuropathy
* Chronic pathology that may interfere with the neurophysiological assessment
* Patient who were given anticoagulation drug therapy, anti-cholinergic drugs, beta-blocker and impossibility to withdraw the treatment before neurophysiological tests

In diabetic patients without chronic cough, another non-inclusion criteria is acute or chronic cough

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2022-06-14 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with small fiber neuropathy | 6 month after inclusion visit
  The primary endpoint is the proportion of patients with small fiber neuropathy between diabetic patients with chronic cough and those without chronic cough (defined by at least 2 abnormal neurophysiological tests).

SECONDARY OUTCOMES:
proportion of patients with abnormal results of the thermotest | 6 month after inclusion visit
  estimate the proportion of patients with abnormal results of the thermotest in each arm (with and without chronic cough)
proportion of patients with pathological results of the sudori-motor response | 6 month after inclusion visit
  estimate the proportion of patients with pathological results of the sudori-motor response in each arm (with and without chronic cough)
the proportion of patients with abnormal results of cardiovascular tests | 6 month after inclusion visit
  estimate the proportion of patients with abnormal results of cardiovascular tests assessing the autonomic nervous system in in each arm (with and without chronic cough)
proportion of patients with abnormal results of laser evoked potentials | 6 month after inclusion visit
  estimate the proportion of patients with abnormal results of laser evoked potentials in each arm (with and without chronic cough)
proportion of patients with abnormal findings of cutaneous biopsy | 6 month after inclusion visit
  estimate the proportion of patients with abnormal findings of cutaneous biopsy in in each arm (with and without chronic cough)
values of Leicester Cough Questionnaire (LCQ) in diabetic patients | 6 month after inclusion visit
  estimate the values of Leicester Cough Questionnaire in diabetic patients with and without chronic cough. The Leicester Cough Questionnaire comprises 19 items and takes 5 to 10 minutes to complete. Each item assesses symptoms, or the impact of symptoms, over the last 2 weeks on a seven-point Likert scale. Scores in three domains (physical, psychological and social) are calculated as a mean for each domain (range 1 to 7). A total score (range 3 to 21) is also calculated by adding the domain scores together. Higher scores indicate better quality of life.
values of the DN4 questionnaire in diabetic patients | 6 month after inclusion visit
  estimate the values of the DN4 questionnaire in diabetic patients with and without chronic cough.
  It allows to estimate the probability of neuropathic pain in a patient, through 4 questions divided into 10 check items. The practitioner questions or examines the patient and completes the questionnaire himself. He notes a response ("yes", "no") to each item. At the end of the questionnaire, he counts the answers and assigns the note 1 for each "yes", and the score 0 for each "no". The sum obtained gives the score of the patient, scored out of 10.

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Guilleminault, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Hôpital Larrey, Toulouse, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chung KF. Chronic 'cough hypersensitivity syndrome': a more precise label for chronic cough. Pulm Pharmacol Ther. 2011 Jun;24(3):267-71. doi: 10.1016/j.pupt.2011.01.012. Epub 2011 Feb 1. PMID 21292019
- [Background] De Santi F, Zoppini G, Locatelli F, Finocchio E, Cappa V, Dauriz M, Verlato G. Type 2 diabetes is associated with an increased prevalence of respiratory symptoms as compared to the general population. BMC Pulm Med. 2017 Jul 17;17(1):101. doi: 10.1186/s12890-017-0443-1. PMID 28716044
- [Background] Pavy-Le Traon A, Fontaine S, Tap G, Guidolin B, Senard JM, Hanaire H. Cardiovascular autonomic neuropathy and other complications in type 1 diabetes. Clin Auton Res. 2010 Jun;20(3):153-60. doi: 10.1007/s10286-010-0062-x. Epub 2010 Mar 31. PMID 20354891
- [Background] Casellini CM, Parson HK, Richardson MS, Nevoret ML, Vinik AI. Sudoscan, a noninvasive tool for detecting diabetic small fiber neuropathy and autonomic dysfunction. Diabetes Technol Ther. 2013 Nov;15(11):948-53. doi: 10.1089/dia.2013.0129. Epub 2013 Jul 27. PMID 23889506